CLINICAL TRIAL: NCT00443287
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Trial of HMR1766 Assessing the Efficacy and Safety of 3 Doses of HMR1766 Versus Placebo With Cilostazol as a Calibrator, Administered for 26 Weeks in Patients With Peripheral Arterial Disease (PAD) Fontaine Stage II
Brief Title: Efficacy and Safety of HMR1766 in Patients With Fontaine Stage II Peripheral Arterial Disease
Acronym: ACCELA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DFI6174; EudraCT : 2006-004275-35
Record Dates: First submitted 2007-03-02; First posted 2007-03-05 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Intermittent Claudication
Keywords: Peripheral; Artery; Disease
MeSH Terms: conditions — Intermittent Claudication; Disease | interventions — 5-chloro-2-(5-chlorothiophene-2-sulfonylamino)-N-(4-(morpholine-4-sulfonyl)phenyl)benzamide; Cilostazol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- 1 (Placebo Comparator)
  Interventions: Drug: placebo
- 2 (Experimental): dose level 1
  Interventions: Drug: ataciguat (HMR1766)
- 3 (Experimental): dose level 2
  Interventions: Drug: ataciguat (HMR1766)
- 4 (Experimental): dose level 3
  Interventions: Drug: ataciguat (HMR1766)
- 5 (Active Comparator)
  Interventions: Drug: cilostazol

INTERVENTIONS:
Drug: ataciguat (HMR1766) — oral administration
  Arms: 2; 3; 4
Drug: placebo — oral administration
  Arms: 1
Drug: cilostazol — oral administration
  Arms: 5

SUMMARY:
The primary objective is to investigate in patients suffering from intermittent claudication due to Fontaine stage II Peripheral Arterial Disease (PAD) whether a 26-week treatment by HMR1766 on top of clopidogrel may result in an improvement of walking capacity, by comparing three doses of HMR1766 to placebo, and calibrating such effect versus cilostazol.

ELIGIBILITY:
Inclusion Criteria:

* Patient with stable symptoms of intermittent claudication of the lower extremities, secondary to chronic occlusive arterial disease from atherosclerosis etiology (symptoms present for 6 months or longer and not significantly changed within the past 3 months)
* Initial claudication distance of 30 to 250 meters at screening constant workload treadmill test
* Confirmation of underlying Peripheral Arterial Disease (PAD) at screening
* Confirmation of symptom stability at randomization based on constant workload treadmill test performance
* The patient must have optimal cardiovascular risk prevention and appropriate management of PAD, including clopidogrel at the dose of 75mg per day, during the study period

Exclusion Criteria:

* Patient participated in investigational clinical trials in the last month prior to screening
* Pregnant or breast-feeding woman or woman without documented double birth control measures for at least 3 months prior to randomization
* Symptoms of PAD before the age of 40 years
* Recent initiations or discontinuation of treatment by vasoactive agents (e.g., pentoxifylline, berprost sodium, papverine, isoxsuprine, nylidrin, cyclandelate, and niacin derivatives). Patients treated by cilostazol within 3 months prior to screening will also be excluded
* Recent lower-extremity surgical or endovascular arterial reconstructions or sympathectomy, or recent deep venous thrombosis
* Recent occurrence of at least one of the following: acute myocardial infarction, unstable angina, coronary artery bypass graft, percutaenous coronary intervention, transient ischemic attack or stroke

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 553 (Actual)
Dates: Start 2007-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Primary efficacy endpoint: percent change in initial claudication distance (ICD) measured at the 26-week treadmill test, compared with ICD measured at baseline | 26 weeks

SECONDARY OUTCOMES:
Secondary efficacy endpoint: percent change in the absolute claudication distance | 26 weeks
Safety endpoints: adverse events | study period

CONTACTS AND LOCATIONS:
Overall Officials: ICD, Study Director — Sanofi
Locations (7):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Midrand, South Africa